CLINICAL TRIAL: NCT01450475
Title: A Randomized Control Trial of Effect of Remote Ischemic Postconditioning on Children Undergoing Cardiac Surgery
Brief Title: Study of Remote Ischemic Postconditioning
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, wangqiang, department of anesthesijology, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: mazuike-18
Record Dates: First submitted 2011-10-09; First posted 2011-10-12 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-07

CONDITIONS: Ischemia; Bypass Complications
MeSH Terms: conditions — Ischemia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Remote ischemic postconditioning (Experimental): At the time of reperfusion, remote ischaemic postconditioning will be induced by inflating a cuff around leg to 100 mmHg for 5 mins followed by 5 mins of reperfusion. This cycle will be repeated 3 times.
  Interventions: Procedure: Remote ischemic postconditioning
- control (No Intervention): A blood cuff was around leg without inflation or deflation.

INTERVENTIONS:
Procedure: Remote ischemic postconditioning — At the time of reperfusion, remote ischaemic postconditioning will be induced by inflating a cuff around leg to 100 mmHg for 5 mins followed by 5 mins of reperfusion. This cycle will be repeated 3 times.
  Other Names: Limb ischemic postconditioning
  Arms: Remote ischemic postconditioning

SUMMARY:
Cardiac surgery is associated with cardiac and cerebral injury because of ischemia/reperfusion in approximately one third of cases. Ischemic preconditioning (IPC), have been shown to reduce the extent of myocardial infarction (MI). As another ischemic conditioning, remote ischemic postconditioning, limits MI size in animal models. The purpose of this study is to evaluate the cardiac and cerebral protective effect of remote ischemic postconditioning in children undergoing cardiac surgery, as a single-center, randomized controlled trial.

DETAILED DESCRIPTION:
Cardiac surgery is associated with Troponin release because of ischemia/reperfusion injury in approximately one third of cases. And I/R injury may also induce cerebral insult, even Postoperative Cognitive Dysfunction (POCD).Transient sublethal episodes of ischemia before a prolonged ischemia/reperfusion injury, known as ischemic preconditioning (IPC), have been shown to reduce the extent of myocardial infarction (MI).And remote ischemic postconditioning(RIPoC), as another ischemic condition, limits MI size in animal models.

However, there are limited outcome to demonstrate protection from RIPoC during cardiac surgery. The purpose of this study is to investigate the cardiac and cerebral protective effect of remote ischemic postconditioning , as a single-center, randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* All Children aged from 0 to 12 who are undergoing open congenital cardiac surgery.

Exclusion Criteria:

* Simple atrial septal defect
* Bidirectional cavopulmonary shunt undergoing Fontan completion
* Chromosomal defects
* Airway or parenchymal lung disease
* Immunodeficiency
* Blood disorder

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2011-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
cTnI,CK-MB concentration | 24h after Remote Ischemic Postconditioning
  The primary outcome is assessing whether cTnI or CK-MB concentration reduce at 24 hours after remote ischemic postconditioning.

SECONDARY OUTCOMES:
NSE，S100β concentration | 24 hours after Remote Ischemic Postconditioning
  The secondary outcome is assessing whether NSE or S100-β concentration reduce at 24 hours after remote ischemic postcondioning.

CONTACTS AND LOCATIONS:
Overall Officials: Wang Qiang, doctor, Study Director — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China